CLINICAL TRIAL: NCT01677221
Title: A Clinical Trial Investigating the Effects of Acleara Needle Insert on Acne Vulgaris
Brief Title: Effects of Acleara Needle Insert on Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theravant Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acleara-01
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Acne Vulgaris
Keywords: acne; inflammatory acne; intense pulsed light
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Acleara Acne Treatment System

SUMMARY:
This prospective, open-label study will be conducted in 15 healthy subjects per clinical site ages 14 or older who meet the inclusion/exclusion criteria. Each subject may have up to 5 lesions treated on the face, chest or back with the Acleara insert. Subjects will receive up to 3 follow up visits and evaluated for improvement in acne lesions and monitored for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >14 years of age
* Subject has mild to moderate acne vulgaris on the face, chest or back.
* Subject has one or more inflammatory acne lesions on face, chest or back.
* Willingness to participate in the study
* Informed consent agreement signed by the subject
* Willingness to follow the treatment schedule and post treatment care requirements
* Willingness to remain on current acne therapy as directed by the Investigator.

Exclusion Criteria:

* Subject has an infection or other dermatologic condition (aside from acne) in the area to be treated
* Subject is immunosuppressed
* Subject is unable to comply with treatment or follow-up visits
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Subject assessment of reduction in acne lesion size | 24-72 hours, 1-2 weeks, 1 month
  Percentage range of lesion reduction

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Charles County Dermatology Associates, White Plains, Maryland
  - Bellaire Dermatology Associates, Bellaire, Texas